CLINICAL TRIAL: NCT07312539
Title: The Influence of Potential Risk Factors on the Long-Term Success of Mineral Trioxide Aggregate Pulpotomy in Primary Teeth
Brief Title: Risk Factors on the Long-Term Success of Mineral Trioxide Aggregate Pulpotomy
Status: Completed | Type: Observational
Sponsor: Sümeyra Akkoç (Other)
Responsible Party: Sponsor-Investigator, Sümeyra Akkoç, Assistant Professor, DDS, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Other Study IDs: 2024/08-27
Record Dates: First submitted 2025-11-29; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Tooth, Deciduous; Pulpotomy; Risk Factors; Mineral Trioxide Aggregate (MTA)
Keywords: Pediatric dentistry; Pulpotomy in primary teeth; Restoration quality; Regression analysis; Mineral Trioxide Aggregate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the long-term results of Mineral Trioxide Aggregate (MTA) pulpotomy in primary molars and the factors that may affect treatment success.

The main question it aims to answer is:

Do clinical, operator and restoration-related factors influence the long-term success of MTA pulpotomy in primary molars?

In this study, children who received MTA pulpotomy treatment were examined at the 24-month follow-up visit, scheduled at the beginning of the study. Two examiners checked the clinical condition of the teeth, and two other examiners reviewed the radiographs without knowing the clinical results.

DETAILED DESCRIPTION:
This cross-sectional observational study was conducted to evaluate the 24-month clinical and radiographic outcomes of Mineral Trioxide Aggregate (MTA) pulpotomy in primary molars and to identify potential risk factors associated with treatment failure. The study included 175 primary molars from 96 children who met the inclusion criteria and were invited to the 24-month follow-up visit scheduled at the beginning of the study. At this visit, two clinical examiners assessed the clinical condition of the teeth, and two radiographic examiners, blinded to the clinical data, evaluated the radiographic outcomes.

Clinical and radiographic findings were scored based on criteria originally established by Zurn and Seale, subsequently adapted by Rajasekharan et al., and recently by Cordell et al. The risk factors that could have influenced treatment failure were also documented, including arch type (maxillary or mandibular), tooth type (first or second primary molar), side (right or left), number of restored surfaces, and restoration quality. Restoration quality was assessed using the modified FDI criteria assessing esthetic, functional, and biological properties.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children
* Complete preoperative clinical and radiographic records available
* No additional treatment performed on the treated tooth after the initial MTA pulpotomy
* Attendance at the 24-month follow-up appointment
* Willingness to participate in the study
* Positive or definitely positive behavior during the clinical examination at the 24-month follow-up visit (Frankl Behavior Rating Scale: + or ++)

Exclusion Criteria:

* Teeth that had exfoliated or received treatment at another center during the follow-up period

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consisted of patients aged 3 to 15 years at the time of treatment, who received pulpotomy treatment using MTA in at least one primary molar between July 1 and November 1, 2022. To evaluate the treatment outcomes and potential risk factors for treatment failure, follow-up appointments were scheduled 24 months after the pulpotomy procedure, and patients were invited to attend at that time in accordance with the order of patient registration.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | Patients were recalled for evaluation at 24 months post-treatment; follow-up was complete when the last enrolled patient attended the 24-month visit.
  Clinical outcome was evaluated at 24 months post-treatment by clinical examination using the standardized criteria defined by Zurn and Seale. Scores of 1-2 were classified as treatment success and scores of 3-4 as treatment failure, and results were reported as the proportion of teeth with clinical success (%).
Radiographic outcome | Patients were recalled for evaluation at 24 months post-treatment; follow-up was complete when the last enrolled patient attended the 24-month visit.
  Radiographic outcome was evaluated at 24 months post-treatment by clinical examination using the standardized criteria defined by Zurn and Seale. Scores of 1-2 were classified as treatment success and scores of 3-4 as treatment failure, and results were reported as the proportion of teeth with clinical success (%).

OTHER OUTCOMES:
Potential risk factors associated with treatment failure | Patients were recalled for evaluation at 24 months post-treatment; follow-up was complete when the last enrolled patient attended the 24-month visit.
  Treatment outcome (success vs failure) was analyzed using binary logistic regression with prespecified predictors including arch type (maxillary/mandibular), tooth type (first/second primary molar), side (right/left), number of restored surfaces, operator, and restoration quality. Results were reported as adjusted odds ratios (ORs) with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Şevval Çakıcı, Assistant Professor, DDS, Principal Investigator — Department of Pediatric Dentistry, Faculty of Dentistry, Kütahya Health Sciences University; Beyza Ecem Alkaç Ekici, Assistant Professor, DDS, Principal Investigator — Department of Pediatric Dentistry, Faculty of Dentistry, Kütahya Health Sciences University; Merve Uluakay, Assistant Professor, DDS, Principal Investigator — Department of Pediatric Dentistry, Faculty of Dentistry, Kütahya Health Sciences University
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Kütahya Health Sciences University, Kütahya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to privacy or ethical restrictions but are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Zurn D, Seale NS. Light-cured calcium hydroxide vs formocresol in human primary molar pulpotomies: a randomized controlled trial. Pediatr Dent. 2008 Jan-Feb;30(1):34-41. PMID 18402097
- [Result] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Result] Kim CH, Bae JS, Kim IH, Song JS, Choi HJ, Kang CM. Prognostic factors for the survival of primary molars following pulpotomy with mineral trioxide aggregate: a retrospective cohort study. Clin Oral Investig. 2021 Apr;25(4):1797-1804. doi: 10.1007/s00784-020-03482-3. Epub 2020 Aug 4. PMID 32754786
- [Result] Yu Y, Hao S, Jin Y, Zhang Q, Wang Y, Zou J. Potential factors affecting the success rate of indirect pulp therapy in primary molars with deep caries: a retrospective study. J Clin Pediatr Dent. 2024 May;48(3):46-51. doi: 10.22514/jocpd.2024.058. Epub 2024 May 3. PMID 38755981
- [Result] An Y, Ferretti M, Bresler R, Pham E, Ferretti GA. Biodentine as a pulpotomy medicament for primary molars: a retrospective chart review. J Clin Pediatr Dent. 2024 Jan;48(1):85-90. doi: 10.22514/jocpd.2024.011. Epub 2024 Jan 3. PMID 38239160